CLINICAL TRIAL: NCT00067509
Title: A Second Chance With Emergency Contraception (ECP): Reducing Unintended Pregnancy
Brief Title: Emergency Contraception (ECP): Reducing Unintended Pregnancies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: HD38515
Record Dates: First submitted 2003-08-21; First posted 2003-08-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-07

CONDITIONS: Contraception; Pregnancy
Keywords: Female
MeSH Terms: interventions — Contraception, Postcoital; Estrogens; Progesterone

INTERVENTIONS:
Drug: emergency contraception (estrogen/progesterone)

SUMMARY:
Emergency contraception is a method of birth control that can be used up to three days after sexual intercourse. Emergency contraceptive pills (ECPs) can be given to a woman before she needs them (advance provision) or when she needs them (emergency provision). This study will compare these two methods of providing ECPs.

DETAILED DESCRIPTION:
ECPs can give women a "second chance" to prevent an unintended pregnancy that might arise because of lack or improper/defective use of contraceptives. By using ECP, a woman can reduce her risk of pregnancy by at least 75%; however, there is little information on what distribution patterns and other factors are most likely to encourage ECP use. This study will compare the use and cost of two ECP distribution patterns: advance provision and emergency provision. It will also identify environmental, situational, and behavioral factors associated with ECP acceptance and use.

Participants in this study will be recruited from four family planning clinics in the Philadelphia area and five family planning clinics in the Pittsburgh area. Participants from the Philadelphia clinics will be given ECPs as part of a regular clinic visit (advance provision); participants from the Pittsburgh clinics will be given ECPs on an emergency basis (emergent provision). Each participant will complete a short intake form and will be issued a pager. Participants will be paged every month over an 18-month period as a reminder to respond to a short automated telephone survey on ECP, contraceptives, and pregnancy status. Approximately half of the participants will be randomly selected to participate in in-depth interviews at study entry and Months 9 and 18. Clinic visit data will augment the surveys to verify use of the clinic and contraceptive method and to develop cost data.

ELIGIBILITY:
Inclusion Criteria

* Patient at a participating clinic

Exclusion Criteria

* Pregnant
* Medical or surgical procedure preventing pregnancy (e.g., tubal ligation, hysterectomy)
* Norplant or IUDs
* Desires to become pregnant

Ages: 15 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1100
Dates: Start 2001-06; Study Completion 2004-05

CONTACTS AND LOCATIONS:
Overall Officials: Paul G Whittaker, D.Phil., Principal Investigator
Locations (2):
- United States (2):
  - Family Planning Council, Philadelphia, Pennsylvania
  - Family Health Council, Pittsburgh, Pennsylvania